CLINICAL TRIAL: NCT02088359
Title: Compare of Effectiveness Cycled Light or Near Darkness on Growth Parameters in Preterm Infants
Status: Completed | Type: Observational
Sponsor: Zekai Tahir Burak Women's Health Research and Education Hospital (Other)
Responsible Party: Principal Investigator, Mehmet Yekta, Zekai Tahir Burak Maternity and Teaching Hospital, Zekai Tahir Burak Women's Health Research and Education Hospital
Other Study IDs: ZTB000123
Record Dates: First submitted 2014-03-07; First posted 2014-03-14 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2012-06

CONDITIONS: Compare of Effectiveness Cycled Light and Near Darkness on Growth in Preterm Infants
Keywords: cycled light, near darkness, growth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Cycled light: Approximately 12 hours of light on and 12 hours of light off.
  Interventions: Other: Cycled light
- Near darkness: Continue near darkness
  Interventions: Other: Continue near darkness

INTERVENTIONS:
Other: Cycled light — We covered the incubator with blanket for darkness approximately 12 hours.
  Groups: Cycled light
Other: Continue near darkness — We covered the incubator with blanket all days.
  Groups: Near darkness

SUMMARY:
Infants are exposed to either continuous bright light continuous near darkness or unstructured combination of the two. The investigators primary objective is to determine the effectiveness cycled light and near darkness on growth in preterm infants.

ELIGIBILITY:
Inclusion Criteria:

* <32 gestational weeks preterm infants

Exclusion Criteria:

* Major congenital anomaly
* Small for gestation age
* Grade III-IV intracranial hemorrhage

Max Age: 24 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Preterm infant (<32 gestational weeks) were enrolled in this study.
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2012-06; Primary Completion 2013-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Effectiveness on growth | 3-12 months
  We recorded infants' weight, height and head circumference measures on day 14, corrected 3 and 6 months.

SECONDARY OUTCOMES:
Feeding | 0-1 month
  We evaluated full enteral feeding time between two groups.
Ventilation support | 0-1 month
  We evaluated duration of supplemental oxygen, nasal continuous positive airway pressure (CPAP) and mechanical ventilation for each groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Zekai Tahir Burak Maternity Teaching Hospital, Ankara, Turkey (Türkiye)

REFERENCES:
- [Derived] Morag I, Xiao YT, Bruschettini M. Cycled light in the intensive care unit for preterm and low birth weight infants. Cochrane Database Syst Rev. 2024 Dec 19;12(12):CD006982. doi: 10.1002/14651858.CD006982.pub5. PMID 39699174